CLINICAL TRIAL: NCT00487045
Title: Prevention and/or Reduction of Hemorrhoids and/or Thrombosed External Hemorrhoids (TEH) Using the HEM-AVERT Perianal Stabilizer Instrument
Brief Title: Prevention and/or Reduction of Hemorrhoids and/or Thrombosed External Hemorrhoids Using the HEM-AVERT Perianal Stabilizer Instrument
Acronym: HEM-AVERT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stetrix, Inc. (Industry)
Collaborators: Baptist Memorial Health Care Corporation (Other)
Responsible Party: David Blurton, CEO of Plexus Biomedical, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB_001
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; Thrombosed External Hemorrhoids (TEH); Reduction; Prevention; Stabilizer Device; Pregnant; Vaginal Birth; Single Birth; Asymptomatic Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Hem-Avert Perianal Stabilizer, single use, disposable, sterile, individually packaged instrument
  Interventions: Device: Hem-Avert Perianal Stabilizer
- 2 (No Intervention)

INTERVENTIONS:
Device: Hem-Avert Perianal Stabilizer — Hem-Avert Perianal Stabilizer, TNP-01L, single-use, disposable, sterile, individually packaged instrument
  Arms: 1

SUMMARY:
This study is being conducted to evaluate an investigational instrument called the HEM-AVERT Perianal Stabilizer and its efficacy in reducing the occurrence or severity of hemorrhoids and thrombosed external hemorrhoids (TEH) which commonly occur during vaginal delivery.

DETAILED DESCRIPTION:
This study is being conducted to evaluate an investigational instrument called the HEM-AVERT™ Perianal Stabilizer and its efficacy in reducing the occurrence or severity of hemorrhoids and thrombosed external hemorrhoids (TEH). Hemorrhoids and TEH are caused by blood pooling in a distended vein and forming a clot, or thrombose, in the outer region of the anus. An anal fissure is a small split or tear in the anal mucosa that may result in painful bowel movements and bleeding. Like hemorrhoids, anal fissures are common in women after childbirth. Lacerations are graded as first, second, third and fourth degree. First and second degree are perineal lacerations and involve the mucosa and perineum and usually heal by themselves. First and second degree lacerations are considered to be a normal occurrence in child birth. Third degree lacerations involve the anal sphincter and fourth degree lacerations involve the sphincter and mucosa of the anus with bowel involvement and usually require surgical repair. Per the product classification that was assigned to this instrument by the FDA, the instrument is both non-invasive and posses a non-significant risk. It is classified as a manual, general instrument with no specific indications, but has a general indication of stabilizing pressure. The purpose of this clinical study is to collect data to support a 510(k) application to obtain the specific indication of preventing the occurrence of hemorrhoids, or reducing the severity of hemorrhoids which often occur during vaginal deliveries. Hemorrhoids and TEH represent common adverse events in vaginal births with reported occurrences ranging from a low of 9% to a high of 34% in the reported literature. Currently no preventative treatment exists. There will be two study groups; an investigational group (subjects receiving the HEM-AVERT™ instrument) and the control group (subjects will not receive the HEM-AVERT™ instrument). The HEM-AVERT™ Perianal Stabilizer is a Class 1, exempt device in accordance with FDA regulation 21 CFR 890.5765. The HEM-AVERT™ is a non-invasive instrument used to provide continuous pressure to the perianal region as a means to help provide support during the labor process. Each HEM-AVERT™ instrument is a single use, disposable, sterile, individually packaged instrument. The HEM-AVERT™ instrument consists of three components: 1) a rigid polymer base manufactured from a medical grade polycarbonate; 2) a centrally located cushioning pad which is composed of a laminate of medical grade polyester non-woven tape and medical grade polyethylene foam tape; and 3) two lateral hook and loop fastener adhesive strips (with liners) ("loop" strips that attach to the mating "hook" [similar to VELCRO®]) which is used to provide the tension needed to keep the instrument firmly in place during delivery. The cushioning pad and adhesive strips are manufactured using materials commonly found in medical instruments and used in medical procedures. All of the materials used to manufacture this instrument meet the available national or international standards specifications as applied to this instrument. This instrument is not to be implanted.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 40 years of age, female and pregnant.
* Subject weighs 130 pounds or greater at time of delivery.
* Subject is scheduled for vaginal delivery.
* Subject is willing and able to comply with the study plan as indicated by understanding and signing the Subject Informed Consent Form.
* Subject's pre-natal examination indicates that this is to be a single birth delivery.
* Subject has no current hemorrhoids or has low grade hemorrhoids.
* Subject's with previous history of hemorrhoids that are visually asymptomatic at time of screening (history) and physical examination are also acceptable
* Subject has no lacerations or anal fissures
* Subject is not a prisoner

Exclusion Criteria:

* Subject is younger than 18 years of age or older than 40 years of age.
* Subject weighs less than 130 pounds at time of delivery.
* Subject has hemorrhoids other than low grade
* Subject has had previous rectal surgery (e.g., hemorrhoidectomy)
* Subject has lacerations or anal fissures
* Subject has a documented allergy to the instrument's materials.
* Subject's scheduled for vaginal delivery with anticipated complications [such as breech presentation]
* Subject is unable to understand and sign the informed consent form.
* Subject is a prisoner.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the success rate and assess the safety and efficacy of the HEM-AVERT™ instrument as a method of reducing the occurrence and/or severity of hemorrhoids and/or Thrombosed External Hemorrhoids (TEH), which commonly occur during vaginal delivery. | Screening(Baseline), Delivery , Follow-up at Discharge (Total = 3 to 4 months)

SECONDARY OUTCOMES:
Grade presence or absence, # present, % of circumference of anus involved and volume of burden of hemorrhoids before & after delivery in both groups. Compare the occurrence of lacerations, anal fissures, and C-Sections in both groups. | Screening(Baseline), Delivery, Follow-up at Discharge (Total = 3 to 4 months)

CONTACTS AND LOCATIONS:
Overall Officials: J. Bradley Stern, M.D., Principal Investigator — Baptist Memorial Health Care Corporation
Locations (3):
- United States (3):
  - Baptist Memorial Hospital-Desoto, Southaven, Mississippi
  - Baptist Memorial Hospital-Tipton, Covington, Tennessee
  - Baptist Women's Hospital, Memphis, Tennessee

REFERENCES:
- [Background] Abramowitz L. et.al. Epidemiology of anal fissures (fissure and thrombosed external hemorrhoid) during pregnancy and post-partum. Gynecxologie Obstetrique Fertilite, 31:546-549, 2003. Abramowitz L. et.al. Anal fissures and thrombosed external hemorrhoids before and after delivery. Dis. Colon Rectum, 45:650-655, 2002. Brown S, Luley J. Maternal health after childbirth: Results of an australian population based survey. British Journal Obstet Gynaecol. 105(2):156-161, 1998. Byrd LM, Hobbiss J, Tasker M. Is it possible to predict or prevent third degree tears? Colorectal Disease. 7(4):311-318, 2005. Gjerdingen DK, Froberg DG, Chaloner KM, McGovern, PM. Changes in women's physical health during first postpartum year. Arch Fam Med. 2:277-283, 1993. Cohen J. Statistical power analysis for the behavioral sciences. Second Edition. Hillsdale NJ: Lawrence Erlbaum Associates,Inc. 1988.